CLINICAL TRIAL: NCT00146757
Title: A Phase II Open-Label Clinical Trial of Recombinant Human Alpha-L-iduronidase (Aldurazyme®) to Evaluate the Safety and Pharmacokinetics in Mucopolysaccharidosis I (MPS I) Patients Less Than 5 Years Old
Brief Title: A Study Evaluating the Safety and Pharmacokinetics of Aldurazyme® (Laronidase) in MPS I Patients Less Than 5 Years Old
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Collaborators: BioMarin/Genzyme LLC (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALID-014-02
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Results first posted 2009-06-16 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-03

CONDITIONS: Mucopolysaccharidosis I; Hurler Syndrome; Hurler-Scheie Syndrome; Scheie Syndrome
MeSH Terms: conditions — Mucopolysaccharidosis I | interventions — Iduronidase

ARMS (2):
- Aldurazyme (rhIDU) 100 U/kg ONLY every week (Experimental): Patients received Aldurazyme (recombinant human alpha-L-iduronidase (rhIDU)) once per week at a dose of 100 Units/kg (approximately 0.58 mg/kg) for up to 52 weeks - labeled dose.
  Interventions: Biological: Aldurazyme (Recombinant Human Alpha-L-Iduronidase)
- Aldurazyme (rhIDU) 100-200 U/kg every week (Experimental): After receiving 100 Units/kg dose of Aldurazyme (rhIDU) for the first 25 weeks, patients enrolling after January 1, 2004 were eligible to receive an increased dose of 200 Units/kg from Week 26 onwards if the patient's urinary glycosaminoglycan (uGAG) levels were >200µg/mg creatinine at Week 22.
  Interventions: Biological: Aldurazyme (Recombinant Human Alpha-L-Iduronidase)

INTERVENTIONS:
Biological: Aldurazyme (Recombinant Human Alpha-L-Iduronidase) — 100 U/kg every week
  Arms: Aldurazyme (rhIDU) 100 U/kg ONLY every week
Biological: Aldurazyme (Recombinant Human Alpha-L-Iduronidase) — 200 U/kg every week (Week 26 onwards)
  Arms: Aldurazyme (rhIDU) 100-200 U/kg every week

SUMMARY:
The main objectives of this study are to evaluate the safety and pharmacokinetics (PK) of enzyme replacement therapy with recombinant human alpha-L-iduronidase [Aldurazyme® (laronidase)] in mucopolysaccharidosis I (MPS I) patients less than 5 years old. Efficacy measurements will also be evaluated in this study.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent is required from the parent(s) or legal guardian(s) prior to any protocol-related procedures being performed. (A separate informed consent will be requested from the parent(s) for their genotyping, which is independent of the inclusion.)
* Be less than 5 years of age at the time of enrollment.
* Have confirmed iduronidase deficiency with a fibroblast or leukocyte alpha-L-iduronidase enzyme activity level of less than 10.0 % of the lower limit of the normal range, or below the detection range of the measuring laboratory.
* Have a clinical diagnosis of MPS I based on genotyping.
* Documentation in his/her medical record that the parent(s) or legal guardian(s) have had counseling or a consultation regarding HSCT in order to assure that the parent(s) or legal guardian(s) are fully informed regarding the risks and benefits of this alternative treatment for patients eligible for the trial and with the severe manifestations of MPS I with neurodegeneration.

Exclusion Criteria:

* The patient is under consideration for or has undergone hematopoietic stem cell transplantation (HSCT).
* The patient has acute hydrocephalus at the time of enrollment.
* The patient has a clinically significant organic disease (with the exception of symptoms relating to MPS I) including: cardiovascular, hepatic, pulmonary, neurologic, or renal disease, other serious intercurrent illness, or extenuating circumstances that, in the opinion of the Investigator, would preclude participation in the trial or potentially decrease survival.
* The patient has received any investigational product within 30 days prior to trial enrollment.
* The patient has known severe hypersensitivity to Aldurazyme® (laronidase) or components of the delivery solution.

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2002-10; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (4):
- Hôpital E. Herriot, Lyon, France
- Johannes Gutenberg Universität, Kinderklinik, Mainz, Germany
- Sophia Children's Hospital, Rotterdam, Netherlands
- Willink Biochemical Genetics Unit Royal Hospital for Children, Manchester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Aldurazyme (rhIDU) 100 U/kg Every Week: Patients received Aldurazyme (recombinant human alpha-L-iduronidase (rhIDU)) once per week at a dose of 100 Units/kg (approximately 0.58 mg/kg) for up to 52 weeks - labeled dose.
Period: Overall Study
Arm/Group | Aldurazyme (rhIDU) 100 U/kg Every Week | Aldurazyme (rhIDU) 100-200 U/kg Every Week
Started | 16 | 4
Completed | 14 | 4
Not Completed | 2 | 0
Not completed — Death | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Arms 1 and 2 Combined
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 2.9 (1.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 18
  Black | 1
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Safety Evaluation
Description: Overall Safety Summary of Adverse Events (AEs) during Treatment Safety assessment was based on the incidence of AE reports.
Time Frame: 52 weeks
Population: The number of participants was determined as adequate to assess the safety of Aldurazyme in young children with mucopolysaccharidosis I (MPS I). The analysis was intent-to-treat.
Measure: Number; unit: participants
Arm/Group | Aldurazyme (rhIDU) 100 U/kg Every Week | Aldurazyme (rhIDU) 100-200 U/kg Every Week
Number analyzed (Participants) | 16 | 4
participants
  Having Adverse Events (AE) | 16 (21.41) | 4 (14.21)
  Having Drug-Related AEs | 5 | 3
  Deaths/Discontinuations Due to AEs | 2 | 0
  Having Serious AEs | 12 | 3
  Having Severe AEs | 5 | 1
  Having Infusion Associated Reactions (IAR): | 4 | 3

2. Primary Outcome: Pharmacokinetics - Area Under the (Plasma Concentration-time) Curve (AUC∞)
Description: AUC∞ is a measure of the total exposure to a drug.
Time Frame: 52 weeks
Population: The analysis was intent-to-treat.
Measure: Mean (Standard Deviation); unit: hours units/milliliters
Arm/Group | Arms 1 and 2 Combined
Number analyzed (Participants) | 20
hours units/milliliters
  Week 1 | 0.577 (0.591)
  Week 13 | 0.418 (0.246)
  Week 26 | 0.92 (0.68)
  Week 52 | 0.94 (0.97)

3. Primary Outcome: Pharmacokinetics - Elimination Half Life (t1/2)
Description: Half-life is the time it takes for the concentration of drug in plasma to decline by 50%.
Time Frame: 52 weeks
Population: The analysis was intent-to-treat.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Arms 1 and 2 Combined
Number analyzed (Participants) | 20
hours
  Week 1 | 1.55 (0.516)
  Week 13 | 0.55 (0.284)
  Week 26 | 0.946 (0.877)
  Week 52 | 1.147 (0.87)

4. Primary Outcome: Pharmacokinetics - Total Plasma Clearance (CL)
Description: CL is volume of the body fluid cleared of the drug per unit of time.
Time Frame: 52 weeks
Population: The analysis was intent-to-treat.
Measure: Mean (Standard Deviation); unit: (milliliters/minute)/kilograms
Arm/Group | Arms 1 and 2 Combined
Number analyzed (Participants) | 20
(milliliters/minute)/kilograms
  Week 1 | 5.73 (3.90)
  Week 13 | 5.33 (2.67)
  Week 26 | 2.97 (1.87)
  Week 52 | 3.20 (2.02)

5. Primary Outcome: Pharmacokinetics - Volume of Distribution (Vz)
Description: Vz is the volume that relates the amount of drug in the body after absorption is complete to the concentration of drug in the plasma.
Time Frame: 52 weeks
Population: The analysis was intent-to-treat.
Measure: Mean (Standard Deviation); unit: liters/kilograms
Arm/Group | Arms 1 and 2 Combined
Number analyzed (Participants) | 20
liters/kilograms
  Week 1 | 0.753 (0.497)
  Week 13 | 0.299 (0.303)
  Week 26 | 0.214 (0.297)
  Week 52 | 0.246 (0.210)

6. Other Pre Specified Outcome: Percent Change From Baseline to Week 52 in Urinary Glycosaminoglycan (uGAG) Level
Description: Percentage change in the concentration of GAG relative to creatinine (ug GAG/mg creatinine) in urine from Baseline to Week 52; A greater decrease in percent change indicates a greater response.
Time Frame: Baseline to 52 weeks
Population: The analysis was intent-to-treat.
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | Aldurazyme (rhIDU) 100 U/kg Every Week | Aldurazyme (rhIDU) 100-200 U/kg Every Week
Number analyzed (Participants) | 12 | 4
Percentage of change | -59.1 (21.41) | -67.7 (14.21)

7. Other Pre Specified Outcome: Percent Change From Baseline to Week 52 in Liver Size (Hepatomegaly)
Description: Percent change in extent of Liver Edge Below Right Costal Margin (BRCM) measured in centimeters from Baseline to Week 52; A greater decrease in percent change indicates a greater response.
Time Frame: Baseline to 52 weeks
Population: The analysis was intent-to-treat.
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | Arms 1 and 2 Combined
Number analyzed (Participants) | 10
Percentage of change | -69.5 (15.34)

8. Other Pre Specified Outcome: Change From Baseline to Week 52 in Apnea/Hypopnea Index (AHI)
Description: Number of absent (apnea) and shallow (hypopnea) breaths per hour of sleep. A greater decrease in events per hour indicates a greater response.
Time Frame: Baseline to 52 weeks
Population: The analysis was intent-to-treat.
Measure: Mean (Standard Deviation); unit: Events per hour
Arm/Group | Arms 1 and 2 Combined
Number analyzed (Participants) | 14
Events per hour | -2.6 (22.27)

9. Other Pre Specified Outcome: Expert Global Assessment of Sleep Study Results at Week 52 Compared With Baseline
Description: Independent experts provided a global assessment for each sleep study visit as well as the degree of clinically meaningful change over the course of the study. Assessment was based on AHI, severity and frequency of oxygen desaturations and sleep quality.
Time Frame: Baseline to 52 weeks
Population: The analysis was intent-to-treat.
Measure: Number; unit: participants
Arm/Group | Arms 1 and 2 Combined
Number analyzed (Participants) | 15
participants
  Marked Improvement | 1
  Moderate Improvement | 3
  Mild Improvement | 1
  No change | 5
  Slight Worsening | 3
  Moderate Worsening | 1
  Marked Worsening | 1

10. Other Pre Specified Outcome: Change From Baseline to Week 52 in Left Ventricular Mass (LVM) Z-Score
Description: Change in LVM Z-scores as measured by echocardiography from Baseline to Week 52. Z-score=number of standard deviations from mean. Z-scores greater than +2 and less than -2 are abnormal. A greater decrease in abnormally high z-score indicates a greater response.
Time Frame: Baseline to 52 weeks
Population: The analysis was intent-to-treat.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Arms 1 and 2 Combined
Number analyzed (Participants) | 17
Units on a scale | -0.9 (1.58)

11. Other Pre Specified Outcome: Change From Baseline to Week 52 in Height
Description: Change in Z-scores for standing height/lying-length-for-age from Baseline to Week 52. Z-score=number of standard deviations from mean. Z-scores greater than +2 and less than -2 are abnormal. A greater decrease in abnormally high z-score indicates a greater response.
Time Frame: Baseline to 52 weeks
Population: The analysis was intent-to-treat.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Arms 1 and 2 Combined
Number analyzed (Participants) | 17
Units on a scale | -0.5 (0.93)

12. Other Pre Specified Outcome: Investigator's Clinical Assessment at Week 52 Compared With Baseline
Description: The Investigator's impression of the patient's overall clinical status at Week 52 compared with Baseline.
Time Frame: Baseline to 52 weeks
Population: The analysis was intent-to-treat.
Measure: Number; unit: participants
Arm/Group | Arms 1 and 2 Combined
Number analyzed (Participants) | 18
participants
  Marked Improvement | 0
  Moderate Improvement | 6
  Mild Improvement | 11
  No Change | 1
  Slight Worsening | 0
  Moderate Worsening | 0
  Marked Worsening | 0

ADVERSE EVENTS:
Description: In the event a single participant has experienced both a serious and a non-serious form of the same adverse event term, the individual has been included in the numerator ("number of affected participants") of both adverse event tables.
Groups:
- Aldurazyme ***Check Title***: Aldurazyme ***check title***
Arm/Group | Aldurazyme ***Check Title***
Serious Adverse Events (participants affected / at risk) | 15/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aldurazyme ***Check Title*** (N=20)
Cardiac failure (Cardiac disorders) | 1
Cyanosis (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Hip dysplasia (Congenital, familial and genetic disorders) | 2
Dental caries (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Umbilical hernia (Gastrointestinal disorders) | 1
Catheter related complication (General disorders) | 1
Pyrexia (General disorders) | 1
Ear infection (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 2
Otitis media (Infections and infestations) | 4
Pharyngitis (Infections and infestations) | 1
Post procedural infection (Infections and infestations) | 1
Respiratory syncytial virus infection (Infections and infestations) | 1
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 1
Postoperative respiratory distress (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 2
Blood pressure increased (Investigations) | 1
Medical observation (Investigations) | 1
Oxygen saturation decreased (Investigations) | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 1
Adenoidal disorder (Respiratory, thoracic and mediastinal disorders) | 1
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 2
Adenotonsillectomy (Surgical and medical procedures) | 1
Catheterisation venous (Surgical and medical procedures) | 1
Central venous catheterisation (Surgical and medical procedures) | 3
Ear tube insertion (Surgical and medical procedures) | 1
Ear tube removal (Surgical and medical procedures) | 1
Poor venous access (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aldurazyme ***Check Title*** (N=20)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 2
Angina pectoris (Cardiac disorders) | 1
Aortic valve disease (Cardiac disorders) | 1
Aortic valve incompetence (Cardiac disorders) | 2
Mitral valve incompetence (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Cerumen impaction (Ear and labyrinth disorders) | 2
Ear congestion (Ear and labyrinth disorders) | 1
Ear pain (Ear and labyrinth disorders) | 4
Ear pruritus (Ear and labyrinth disorders) | 1
Otorrhoea (Ear and labyrinth disorders) | 10
Conjunctivitis (Eye disorders) | 3
Eye discharge (Eye disorders) | 1
Lacrimation increased (Eye disorders) | 1
Ocular hypertension (Eye disorders) | 1
Strabismus (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 17
Faecal incontinence (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Lip haematoma (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Retching (Gastrointestinal disorders) | 1
Teething (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 2
Umbilical hernia (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 14
Adverse drug reaction (General disorders) | 1
Catheter related complication (General disorders) | 1
Catheter site discharge (General disorders) | 1
Catheter site swelling (General disorders) | 4
Chills (General disorders) | 4
Crepitations (General disorders) | 1
Cyst (General disorders) | 1
Facial pain (General disorders) | 1
Fatigue (General disorders) | 2
Feeling hot (General disorders) | 2
Gait disturbance (General disorders) | 1
Inflammation (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 20
Abscess (Infections and infestations) | 1
Bacterial disease carrier (Infections and infestations) | 1
Bacterial infection (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 7
Candida nappy rash (Infections and infestations) | 1
Conjunctivitis infective (Infections and infestations) | 1
Ear infection (Infections and infestations) | 5
Eye infection (Infections and infestations) | 2
Fungal infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 6
Gingival abscess (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 8
Oral candidiasis (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Otitis externa (Infections and infestations) | 1
Otitis media (Infections and infestations) | 2
Paronychia (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 2
Rhinitis (Infections and infestations) | 11
Rubella (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 1
Varicella (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Ear injury (Injury, poisoning and procedural complications) | 1
Excoriation (Injury, poisoning and procedural complications) | 1
Face injury (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 3
Gingival injury (Injury, poisoning and procedural complications) | 1
Head injury (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Mouth injury (Injury, poisoning and procedural complications) | 2
Procedural pain (Injury, poisoning and procedural complications) | 1
Skin laceration (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 2
Bacterial culture positive (Investigations) | 1
Blood iron decreased (Investigations) | 3
Blood pressure decreased (Investigations) | 1
Blood pressure increased (Investigations) | 1
Body temperature increased (Investigations) | 1
Breath sounds abnormal (Investigations) | 1
Cardiac murmur (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Heart rate increased (Investigations) | 1
Lymph node palpable (Investigations) | 1
Oxygen saturation decreased (Investigations) | 3
Platelet count increased (Investigations) | 1
Urine analysis abnormal (Investigations) | 1
White blood cell count increased (Investigations) | 1
Fluid intake reduced (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Arthropathy (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Head discomfort (Nervous system disorders) | 1
Headache (Nervous system disorders) | 3
Hemiparesis (Nervous system disorders) | 1
Hyperreflexia (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 3
Listless (Psychiatric disorders) | 1
Restlessness (Psychiatric disorders) | 2
Self-induced vomiting (Psychiatric disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Pruritus genital (Reproductive system and breast disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 17
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 12
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 2
Heat rash (Skin and subcutaneous tissue disorders) | 2
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 10
Rash macular (Skin and subcutaneous tissue disorders) | 2
Swelling face (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Haematoma (Vascular disorders) | 3
Hypertension (Vascular disorders) | 1
Pallor (Vascular disorders) | 1
Vein disorder (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Due to the rarity of the disease, this study is limited by its small sample size and lack of a control group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In multi-site studies, PI can publish after Genzyme publishes or 18 months after study completion. PI gives Genzyme a draft 60 days before publication. Genzyme can ask that confidential information be removed, and can defer publication another 60 days upon notifying PI that it will file a patent application on inventions contained in the draft.